CLINICAL TRIAL: NCT01237899
Title: Study of the Safety, Tolerability, Pharmacokinetics and Effect on Renal Potassium Clearance After Multiple Oral Dosing of LY2623091 in Healthy Volunteers
Brief Title: Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics and Effect on Renal Potassium Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 14121; I4M-MC-MRAB (Other: Eli Lilly)
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney; Renal
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 mg LY2623091 (Experimental): Daily by mouth for 7 days.
  Interventions: Drug: LY2623091
- 10 mg LY2623091 (Experimental): Daily by mouth for 7 days.
  Interventions: Drug: LY2623091
- 25 mg LY2623091 (Experimental): The anticipated dose of LY2623091 was revised down from the original proposed dose level of 100 mg based on safety and tolerability data. The 25 mg LY2623091 was administered daily by mouth for 7 days.
  Interventions: Drug: LY2623091
- 0.3 mg LY2623091 (Experimental): The anticipated dose of LY2623091 was revised down from the original proposed dose level of up to 200 mg. The 0.3 mg LY2623091 was determined based on an interim analysis after the third dose level and was administered daily by mouth for 7 days.
  Interventions: Drug: LY2623091
- Placebo (Placebo Comparator): Daily by mouth for 7 days.
  Interventions: Drug: Placebo
- 50 mg Eplerenone (Active Comparator): Daily by mouth for 7 days.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: LY2623091 — Administered orally.
  Arms: 0.3 mg LY2623091; 1 mg LY2623091; 10 mg LY2623091; 25 mg LY2623091
Drug: Placebo — Administered orally.
  Arms: Placebo
Drug: Eplerenone — Administered orally.
  Arms: 50 mg Eplerenone

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of LY2623091 after multiple oral dosing in healthy men and women of non-childbearing potential. Two cohorts of 16 subjects will participate in 2 dosing periods. Treatment assignment will be double-blind for LY2623091 and placebo (negative control), and open label for eplerenone (positive control).

ELIGIBILITY:
Inclusion Criteria:

* Are healthy men and women of non-childbearing potential as determined by medical history and physical examination.

  * Male subjects: Non-vasectomized male subjects must agree to use 2 medically accepted methods of contraception with all sexual partners during the study and for 90 days following the final dosing.
  * Female subjects: Female subjects must be of non-childbearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy or tubal ligation) or menopause. They should be a minimum of 12 months without a menstrual period. Peri-menopausal women who are 6 months without a menstrual period.
* Have given written informed consent prior to any study-specific procedures.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow site-specific study procedures.
* Have a body mass index (BMI) of between 19 and 32.5 kilograms per square meter (kg/m^2).
* Have clinical laboratory test results within the normal reference range for the population or study site, or test results with acceptable deviations that are judged by the Investigator not to be clinically significant.
* Have venous access sufficient to allow blood sampling per the protocol.
* Have serum potassium levels within the normal range.
* Are nonsmokers or smokers of less than or equal to 10 cigarettes per day.

Exclusion Criteria:

* Are currently enrolled in, or have discontinued, within 60 days inclusive, a clinical trial involving an investigational drug, device or an off-label use of an approved drug, or are concurrently enrolled in any other type of medical research judged to be scientifically or medically incompatible with this study. Subjects who meet any of these criteria may be enrolled in this study but they cannot be dosed until at least 60 days following the last day of the previous investigational trial.
* Have previously completed or withdrawn from this study or any other study investigating LY2623091.
* Have a history or presence of medical illness including but not limited to any cardiovascular, hepatic, respiratory, hematological, endocrine or neurological disease, or any clinically significant laboratory abnormality that is of a serious medical problem that would preclude study participation.
* Have an abnormality in the 12-lead electrocardiogram (ECG), which increases the risks associated with participation in the study.
* Are unwilling or unable to comply with the use of an electronic data capture system.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody or hepatitis B and/or positive hepatitis B surface antigen.
* Use and/or intend to use any medication for a medical condition that is not compatible with Inclusion Criterion. For medications that may be used in "healthy" subjects (example given: preventative and/or naturopathic agents, temporary symptom-relieving medications, and so forth) the following constraints must be observed:

  * No use of vasoactive drugs (example given: diuretics, antihypertensive agents, phosphodiesterase inhibitors, erectile dysfunction medications, nasal decongestants, et cetera) or systemic glucocorticoids within 7 days of first dosing and/or anticipated use during the study.
  * No use of acetaminophen/paracetamol or non-steroidal anti-inflammatory drugs (NSAIDs) within 24 hours of first dosing and/or anticipated use during the study. Aspirin may not be used at doses greater than 100 milligrams per day (mg/day) within 7days of first dosing and/or anticipated use during the study.
  * No use of herbal or nutritional products within 7 days of first dosing and/or anticipated use during the study.
* Have donated blood of more than 50 milliliters (mL) within the last 60 days.
* Have an average weekly alcohol intake that exceeds 21 units per week and/or subjects unwilling to stop alcohol within 48 hours of study enrollment and for the duration of the study.
* Have an abnormally high blood pressure (supine or standing) defined as diastolic blood pressure greater than 95 millimeters of mercury (mmHg) and /or systolic blood pressure greater than 150 mmHg, confirmed by at least 1 repeat measurement.
* Have serum potassium greater than the upper limit of normal.
* Regularly use known drugs of abuse or show positive findings for such use on urinary drug screening.
* Consumption of natural licorice and/or natural licorice-containing products and/or grapefruit and/or grapefruit juice within 7 days of first dosing and/or anticipated consumption during the study.
* Consumption of methylxanthine-containing beverages and/or foods (example: coffee, tea, caffeinated soft drinks, chocolate) within 4 days of first dosing and/or anticipated consumption during the study.
* Are unwilling to abstain from salt-substitutes containing potassium for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg LY2623091 First Then 25 mg LY2623091: 1 mg LY2623091 daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 25 mg LY2623091 daily by mouth for 7 days.
- 1 mg LY2623091 First Then Placebo: 1 mg LY2623091 daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving placebo daily by mouth for 7 days.
- 1 mg LY2623091 First Then 50 mg Eplerenone: 1 mg LY2623091 daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 50 mg eplerenone daily by mouth for 7 days.
- 50 mg Eplerenone First Then 25 mg LY2623091: 50 mg eplerenone daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 25 mg LY2623091 daily by mouth for 7 days.
- 50 mg Eplerenone First Then Placebo: 50 mg eplerenone daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving placebo daily by mouth for 7 days.
- Placebo First Then 25 mg LY2623091: Placebo daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 25 mg LY2623091 daily by mouth for 7 days.
- 10 mg LY2623091 First Then 0.3 mg LY2623091: 10 mg LY2623091 daily by mouth for 7 days, followed by a minimum 7-day washout period before 0.3 mg LY2623091 daily by mouth for 7 days.
- 10 mg LY2623091 First Then Placebo: 10 mg LY2623091 daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving placebo daily by mouth for 7 days.
- 10 mg LY2623091 First Then 50 mg Eplerenone: 10 mg LY2623091 daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 50 mg eplerenone daily by mouth for 7 days.
- 50 mg Eplerenone First Then 0.3 mg LY2623091: 50 mg eplerenone daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 0.3 mg LY2623091 daily by mouth for 7 days.
- Placebo Then 0.3 mg LY2623091: Placebo daily by mouth for 7 days, followed by a minimum 7-day washout period before receiving 0.3 mg LY2623091 daily by mouth for 7 days.
Period: First Dosing Period
Arm/Group | 1 mg LY2623091 First Then 25 mg LY2623091 | 1 mg LY2623091 First Then Placebo | 1 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 25 mg LY2623091 | 50 mg Eplerenone First Then Placebo | Placebo First Then 25 mg LY2623091 | 10 mg LY2623091 First Then 0.3 mg LY2623091 | 10 mg LY2623091 First Then Placebo | 10 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 0.3 mg LY2623091 | Placebo Then 0.3 mg LY2623091
Started | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4
Completed | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of at Least 7 Days
Arm/Group | 1 mg LY2623091 First Then 25 mg LY2623091 | 1 mg LY2623091 First Then Placebo | 1 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 25 mg LY2623091 | 50 mg Eplerenone First Then Placebo | Placebo First Then 25 mg LY2623091 | 10 mg LY2623091 First Then 0.3 mg LY2623091 | 10 mg LY2623091 First Then Placebo | 10 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 0.3 mg LY2623091 | Placebo Then 0.3 mg LY2623091
Started | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4
Completed | 1 | 3 | 3 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Dosing Period
Arm/Group | 1 mg LY2623091 First Then 25 mg LY2623091 | 1 mg LY2623091 First Then Placebo | 1 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 25 mg LY2623091 | 50 mg Eplerenone First Then Placebo | Placebo First Then 25 mg LY2623091 | 10 mg LY2623091 First Then 0.3 mg LY2623091 | 10 mg LY2623091 First Then Placebo | 10 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 0.3 mg LY2623091 | Placebo Then 0.3 mg LY2623091
Started | 1 | 3 | 3 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4
Completed | 1 | 3 | 3 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg LY2623091 First Then 25 mg LY2623091 | 1 mg LY2623091 First Then Placebo | 1 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 25 mg LY2623091 | 50 mg Eplerenone First Then Placebo | Placebo First Then 25 mg LY2623091 | 10 mg LY2623091 First Then 0.3 mg LY2623091 | 10 mg LY2623091 First Then Placebo | 10 mg LY2623091 First Then 50 mg Eplerenone | 50 mg Eplerenone First Then 0.3 mg LY2623091 | Placebo Then 0.3 mg LY2623091 | Total
Number analyzed (Participants) | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3
  Male | 1 | 2 | 4 | 3 | 2 | 2 | 1 | 3 | 4 | 3 | 4 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  White | 1 | 2 | 4 | 3 | 2 | 4 | 1 | 2 | 4 | 3 | 4 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 1 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 4 | 3 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects (Adverse Events)
Description: A summary of serious adverse events and other nonserious adverse events are located in the Reported Adverse Event section.
Time Frame: Baseline through 7 days for each treatment period
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 0.3 mg LY2623091; 1 mg LY2623091; 10 mg LY2623091; 25 mg LY2623091; 50 mg Eplerenone: Daily by mouth for 7 days.
Arm/Group | Placebo | 0.3 mg LY2623091 | 1 mg LY2623091 | 10 mg LY2623091 | 25 mg LY2623091 | 50 mg Eplerenone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 15
Participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Nonserious Adverse Events | 6 | 2 | 5 | 4 | 6 | 9

2. Secondary Outcome: Pharmacodynamics: Serum to Urine Potassium Area Under the Concentration-Time Curve (AUC) Standardized for Urinary Excretion at Day 7
Description: A measure of the renal clearance of the potassium ion (K+). The Least Squares (LS) Mean value was adjusted for pre-challenge renal K+ clearance.
Time Frame: Day 7: 24 Hour (hr), 48hr and 72hr Postdose
Population: All participants who received at least 1 dose of study drug and for whom the data are considered sufficient and interpretable.
Measure: Least Squares Mean (95% Confidence Interval); unit: liter per hour (L/h)
Arm/Group | Placebo | 0.3 mg LY2623091 | 1 mg LY2623091 | 10 mg LY2623091 | 25 mg LY2623091 | 50 mg Eplerenone
Number analyzed (Participants) | 16 | 8 | 8 | 7 | 6 | 15
liter per hour (L/h) | 2.098 [1.930 to 2.281] | 1.940 [1.748 to 2.153] | 1.981 [1.781 to 2.204] | 1.788 [1.602 to 1.995] | 1.551 [1.383 to 1.739] | 1.838 [1.687 to 2.002]

3. Secondary Outcome: Pharmacokinetics of LY2623091: Maximal Concentration (Cmax) at Day 6
Description: Cmax estimated for LY2623091.
Time Frame: Day 6: Predose,1hr, 2hr, 3hr, 4hr, 8hr and 12 hr Postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.3 mg LY2623091 | 1 mg LY2623091 | 10 mg LY2623091 | 25 mg LY2623091
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanograms per milliliter (ng/mL) | 7.57 (0.776) | 27.5 (5.19) | 324 (55.2) | 812 (106)

4. Secondary Outcome: Pharmacokinetics LY2623091: Area Under the Concentration-Time Curve (AUC) at Day 6
Description: AUC from time 0, extrapolated to infinity, estimated for LY2623091.
Time Frame: Day 6: Predose,1hr, 2hr, 3hr, 4hr, 8hr and 12 hr Postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (µg*h/mL)
Arm/Group | 0.3 mg LY2623091 | 1 mg LY2623091 | 10 mg LY2623091 | 25 mg LY2623091
Number analyzed (Participants) | 8 | 8 | 8 | 8
microgram*hour per milliliter (µg*h/mL) | 0.123 (0.0141) | 0.444 (0.0741) | 5.50 (1.08) | 13.7 (2.37)

ADVERSE EVENTS:
Arm/Group | Placebo | 0.3 mg LY2623091 | 1 mg LY2623091 | 10 mg LY2623091 | 25 mg LY2623091 | 50 mg Eplerenone
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8 | 0/15
Other Adverse Events (participants affected / at risk) | 6/16 | 2/8 | 5/8 | 4/8 | 6/8 | 9/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | 0.3 mg LY2623091 (N=8) | 1 mg LY2623091 (N=8) | 10 mg LY2623091 (N=8) | 25 mg LY2623091 (N=8) | 50 mg Eplerenone (N=15)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vessel puncture site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (6)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days